CLINICAL TRIAL: NCT04794751
Title: Evaluation of Investigational Daily Disposable Multifocal Contact Lenses Produced With Different Manufacturing Processes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-6418
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Results first posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-05

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- senofilcon A C3/delefilcon A/delefilcon A (Experimental): Subjects randomized to this arm will wear the senofilcon A C3 lens during period 1 and the delefilcon A lens during period 2 and period 3
  Interventions: Device: JJVC Investigational Multifocal Contact Lens; Device: Dailies Total 1® Multifocal Contact Lens
- delefilcon A /senofilcon A C3/senofilcon A C3 (Experimental): Subjects randomized to this arm will wear the delefilcon A lens during period 1 and the senofilcon A C3 lens during period 2 and period 3
  Interventions: Device: JJVC Investigational Multifocal Contact Lens; Device: Dailies Total 1® Multifocal Contact Lens

INTERVENTIONS:
Device: JJVC Investigational Multifocal Contact Lens — senofilcon A C3
  Other Names: Test
Device: Dailies Total 1® Multifocal Contact Lens — delefilcon A
  Other Names: Control

SUMMARY:
This is a single-masked, 2×3 crossover, randomized, dispensing clinical trial to evaluate the visual performance and subjective responses of the JJVC Investigational Contact Lens.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all the following criteria to be enrolled in the study:

  1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
  2. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
  3. The subject must be at least 40 years of age and not greater than 70 years of age at the time of consent.
  4. Subjects must own a wearable pair of spectacles if required for their distance vision.
  5. The subject must be an adapted soft contact lens wearer in both eyes (i.e. worn lenses a minimum of 2 days per week for at least 6 hours per wear day, for 1 month or more duration).
  6. The subject must either already be wearing a presbyopic contact lens correction (e.g., reading spectacles over contact lenses, multifocal or monovision contact lenses, etc.) or, if not respond positively to at least one symptom on the "Presbyopic Symptoms Questionnaire" (Appendix E).
  7. The subject's distance spherical equivalent refraction must be in the range of +1.25 D to +3.75 D in each eye.
  8. The subject's refractive cylinder must be ≤0.75 D in each eye.
  9. The subject's ADD power must be in the range of +0.75 D to +2.50 D.
  10. The subject must have distance best corrected visual acuity of 20/20-3 or better in each eye.

      Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Currently pregnant or lactating.
  2. Any active or ongoing ocular or systemic allergies that may interfere with contact lens wear.
  3. Any active or ongoing systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear. This may include, but not be limited to, diabetes, hyperthyroidism, Sjögren's syndrome, xerophthalmia, acne rosacea, Stevens-Johnson syndrome, and immunosuppressive diseases or any infectious diseases (e.g. hepatitis, tuberculosis).
  4. Any previous, or planned, ocular or intraocular surgery (e.g. radial keratotomy, PRK, LASIK, lid procedures, cataract surgery, retinal surgery, etc.).
  5. A history of amblyopia, strabismus or binocular vision abnormality.
  6. Use of any of the following medications within 1 week prior to enrollment: oral retinoid, oral tetracyclines, anticholinergics, oral phenothiazines, oral/inhaled corticosteroids. See Table 9.1 for further examples.
  7. Use of any ocular medication, with the exception of rewetting drops.
  8. History of herpetic keratitis.
  9. History of irregular cornea.
  10. History of pathological dry eye.
  11. Participation in any contact lens or lens care product clinical trial within 30 days prior to study enrollment.
  12. Employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
  13. Any known hypersensitivity or allergic reaction to non-preserved rewetting drop solutions or sodium fluorescein.
  14. Clinically significant (Grade 3 or greater) corneal edema, corneal vascularization, corneal staining, tarsal abnormalities or bulbar injection, or any other corneal or ocular abnormalities which would contraindicate contact lens wear.
  15. Entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions.
  16. Any current ocular infection or inflammation.
  17. Any current ocular abnormality that may interfere with contact lens wear.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2021-03-13 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (7):
- United States (7):
  - VRC-East, Jacksonville, Florida
  - St. Johns Eye Associates, PA, Saint Augustine, Florida
  - Advanced Eyecare, Raytown, Missouri
  - Spectrum Eyecare, Jamestown, New York
  - Sacco Eye Group, Vestal, New York
  - ProCare Vision Centers, Granville, Ohio
  - Tyler Eye Associates, Tyler, Texas

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In total, 78 subject were enrolled in this study. Of those enrolled, 75 subjects were dispensed at least one study lens while 3 subjects failed to meet all eligibility criteria. Of those who were assigned and administered a test article, 64 subjects completed the study while 11 subjects were discontinued.
Groups:
- Delefilcon A/Senofilcon A C3/Senofilcon A C3: Subjects randomized to this sequence received the delefilcon A lens during the first period and then received the senofilcon A C3 lenses during the second and third periods.
- Senofilcon A C3/Delefilcon A/Delefilcon A: Subjects randomized to this sequence received the senofilcon A C3 lens during the first period and then received the delefilcon A lenses during the second and third periods.
Period: Period 1
Arm/Group | Delefilcon A/Senofilcon A C3/Senofilcon A C3 | Senofilcon A C3/Delefilcon A/Delefilcon A
Started | 38 | 37
Completed | 36 | 32
Not Completed | 2 | 5
Not completed — incorrect fitting guide was used to fit subject | 2 | 1
Not completed — Subject no longer meets eligibility criteria | 0 | 1
Not completed — Protocol Violation | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Period: Period 2
Arm/Group | Delefilcon A/Senofilcon A C3/Senofilcon A C3 | Senofilcon A C3/Delefilcon A/Delefilcon A
Started | 36 | 32
Completed | 35 | 29
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — incorrect fitting guide was used to fit subject | 0 | 2
Not completed — Protocol Violation | 1 | 0
Period: Period 3
Arm/Group | Delefilcon A/Senofilcon A C3/Senofilcon A C3 | Senofilcon A C3/Delefilcon A/Delefilcon A
Started | 35 | 29
Completed | 35 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects dispensed a study lens.
Groups:
- Dispensed Subjects: All subjects dispensed a study lens.
Arm/Group | Dispensed Subjects
Number analyzed (Participants) | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (6.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 15
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 4
  Native Hawaiian or Other Pacific Islander | 2
  White | 69
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 75

OUTCOME MEASURES:

1. Primary Outcome: Visual Performance (logMAR)
Description: Binocular visual performance on logMAR (Logarithm of Minimal Angle of Resolution) scale was evaluated at distance (4 m), intermediate (64 cm) and near (40 cm) under high luminance high contrast lighting conditions using ETDRS (Early Treatment Diabetic Retinopathy Study) charts. The room illuminance was required to be between 7.3 and 7.9 EV (394-597 lux). For Distance (4 m), the acceptable range for the chart luminance was 10.5-10.7 EV (181-208 cd/m2). For Intermediate (64cm) and Near (40cm), the cceptable range for the chart luminance 10.8-11.1 EV (223-274 cd/m2). Letter-by-letter results calculated the visual performance score for each chart read. logMAR scores closer to zero, or below zero, indicate a better visual acuity. A logMAR visual performance score of 0.0 is equivalent to Snellen visual acuity of 20/20. The average score was reported for each lens.
Time Frame: 1-Week Follow-up
Population: Subjects that completed all study visits, without a major protocol deviation impacting a primary or secondary endpoint.
Measure: Mean (Standard Deviation); unit: logMAR
Groups:
- Senofilcon A C3: Subjects that wore the Test lens in either of the three study periods.
- Delefilcon A: Subjects that wore the Control lens in either of the three study periods.
Arm/Group | Senofilcon A C3 | Delefilcon A
Number analyzed (Participants) | 64 | 64
logMAR
  Distance (4m) | -0.08 (0.068) | -0.06 (0.081)
  Intermediate (64cm) | -0.01 (0.096) | 0.00 (0.090)
  Near (40cm) | 0.10 (0.094) | 0.09 (0.089)
Statistical Analysis 1: Comparison: Senofilcon A C3 vs Delefilcon A; Distance (4m); Test type: Non-Inferiority — Non-Inferiority was declared if the upper limit of the 95% confidence interval of the LSM difference between the Test and Control was below 0.05 logMAR; Linear Mixed Model; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; least-square mean difference = -0.018, 95% CI 2-sided [-0.039 to 0.002], Standard Error of Mean 0.0106 — LS Mean difference was calculated as Test minus Control
Statistical Analysis 2: Comparison: Senofilcon A C3 vs Delefilcon A; Intermediate (64cm); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Linear Mixed Model; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; least-square mean difference = -0.007, 95% CI 2-sided [-0.032 to 0.018], Standard Error of Mean 0.0127 — LS Mean difference was calculated as Test minus Control
Statistical Analysis 3: Comparison: Senofilcon A C3 vs Delefilcon A; Near (40cm); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Linear Mixed Model; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; least-square mean difference = -0.010, 95% CI 2-sided [-0.034 to 0.015], Standard Error of Mean 0.0124 — LS Mean difference was calculated as Test minus Control

2. Secondary Outcome: CLUE Vision
Description: Subjective vision was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. The average CLUE vision score for each lens type was reported.
Time Frame: 1-Week Follow-up
Population: Subjects that completed all study visits, without a major protocol deviation impacting a primary or secondary endpoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Senofilcon A C3 | Delefilcon A
Number analyzed (Participants) | 64 | 64
units on a scale | 55.34 (20.468) | 55.50 (20.422)
Statistical Analysis 1: Comparison: Senofilcon A C3 vs Delefilcon A; Test type: Non-Inferiority — Non-inferiority was declared if the lower limit of the 95% confidence interval for the least-square mean difference was greater than -5; Linear Mixed Model; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; least-square mean difference = 0.1, 95% CI 2-sided [-4.6 to 4.8], Standard Error of Mean 2.34 — LS Mean difference was calculated as Test minus Control

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study; approximately 22-32 days per subject.
Arm/Group | Senofilcon A C3 | Delefilcon A
All-Cause Mortality (participants affected / at risk) | 0/73 | 0/70
Serious Adverse Events (participants affected / at risk) | 0/73 | 0/70
Other Adverse Events (participants affected / at risk) | 0/73 | 0/70

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-10): https://cdn.clinicaltrials.gov/large-docs/51/NCT04794751/Prot_SAP_000.pdf